CLINICAL TRIAL: NCT06589544
Title: Cost-effectiveness of Transcranial Magnetic Stimulation and Virtual Reality Based Cognitive Remediation on Depressive Symptoms Among Cancer Patients: a Three-arm Randomized Clinical Trial.
Brief Title: Non-pharmacological Care for Depression in Cancer Patients Using VR and TMS
Acronym: INCEPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: University Hospital of Cagliari (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 199/2023/Disp/AUSLFe PNRR onco
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Depressive Symptoms; Quality of Life; Cognitive Impairment
Keywords: Depression; Cognitive functions; Quality of Life; Cancer; Virtual reality; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Neoplasms | interventions — Therapeutics; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality-based Cognitive Remediation (VR-COG) (Experimental): Virtual Reality-based Cognitive Remediation (VR-COG) + Treatment as usual (TAU)
  The "VSail 3D" experimental protocol includes scenarios (virtual environments) dedicated to the sport of sailing. It is based on the software CEREBRUM-VELA (Idego-Promind, srl, Rome, Italy).
  Frequency: 24 sessions, 2 times a week, for 12 consecutive weeks. The duration of each session is 50 minutes.
  Interventions: Device: Virtual Reality-based Cognitive Remediation (VR-COG) + Treatment as Usual (TAU)
- Repetitive transcranial magnetic stimulation (rTMS) (Experimental): Repetitive transcranial magnetic stimulation (rTMS) + Treatment as usual (TAU)
  rTMS group will receive active rTMS using the MagVenture MagPro X100 System (MagVenture A/S, Denmark) equipped with a MagVenture Cool-B65 A/P double-faced coil and a neuronavigation system (Localite GmbH, Sankt Augustin, Germany).
  Frequency: 24 sessions, 2 times a week, for 12 consecutive weeks. The duration of each session is 60 minutes.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS) + Treatment as usual (TAU)
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual (TAU)
  The path, following the guidelines of the Italian Association of Medical Oncology (AIOM-SIPO: https://www.aiom.it), includes an initial psychiatric visit and eventual pharmacological therapy with psychiatric follow-up plus psychological counseling.
  Frequency: 12 weeks. Each counseling session lasts 45-50 minutes, and will be conducted on a monthly basis.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Device: Virtual Reality-based Cognitive Remediation (VR-COG) + Treatment as Usual (TAU) — The "CEREBRUM-VELA" virtual reality software is made up of exercises designed to train different cognitive functions (i.e.: executive functions, motor ability, language). The different degrees of difficulty are designed to adapt to the user's functional diagnosis. Each session, after an initial part of welcome, psychoeducation and orientation to the instrument, involves alternating virtual reality exercises, positive and corrective feedback and suggestions of practical homework that the individual should try to do during his day.
  Treatment as usual (TAU) The path, following the guidelines of the Italian Association of Medical Oncology (AIOM-SIPO: https:// www.aiom.it), includes an initial psychiatric visit aimed at assessing the presence of psychopathological conditions that may necessitate pharmacological therapy (antidepressants, hypnotic-sedatives) and subsequent psychiatric follow-up. The treatment also involves psychological counseling (monthly sessions).
  Arms: Virtual Reality-based Cognitive Remediation (VR-COG)
Device: Repetitive transcranial magnetic stimulation (rTMS) + Treatment as usual (TAU) — Active rTMS stimulation will be delivered at 90% of the resting Motor Threshold (rMT), adjusted for the depth of the fcMRI-identified target. Personalized targets created for each individual will be located at various cortical depths. For safety reasons, the stimulation intensity will never exceed 120% of the rTMS.
  Treatment as usual (TAU) The path, following the guidelines of the Italian Association of Medical Oncology (AIOM-SIPO: https:// www.aiom.it), includes an initial psychiatric visit aimed at assessing the presence of psychopathological conditions that may necessitate pharmacological therapy (antidepressants, hypnotic-sedatives) and subsequent psychiatric follow-up. The treatment also involves psychological counseling (monthly sessions).
  Arms: Repetitive transcranial magnetic stimulation (rTMS)
Other: Treatment as Usual (TAU) — Treatment as usual (TAU) The path, following the guidelines of the Italian Association of Medical Oncology (AIOM-SIPO: https:// www.aiom.it), includes an initial psychiatric visit aimed at assessing the presence of psychopathological conditions that may necessitate pharmacological therapy (antidepressants, hypnotic-sedatives) and subsequent psychiatric follow-up. The treatment also involves psychological counseling (monthly sessions).
  Arms: Treatment as Usual (TAU)

SUMMARY:
Despite its significant impact on individuals and healthcare systems, substantial gaps remain in the clinical and rehabilitative management of depression in oncology patients.

Depression in cancer patients is often under-recognized and untreated, and screening tools and structured healthcare pathways are lacking. Even when depression is identified in oncology patients, evidence of effective treatments is limited. There are no specific guidelines for psychotropic drug use in cancer patients, and antidepressant efficacy is uncertain despite their frequent use.

Emerging strategies like transcranial magnetic stimulation and cognitive rehabilitation show promising findings. However, the cost-effectiveness of therapeutic strategies is understudied.

Repetitive transcranial magnetic stimulation (rTMS) is already used for the treatment and relapse prevention of depression both as monotherapy and as an add-on to antidepressant pharmacotherapy, and it appears effective in improving cognitive performance. However, it has not yet been applied to treat depressive disorders in oncology patients.

Virtual reality-based cognitive behavioral intervention (VR-COG) is designed to improve cognitive functioning, a central feature of depression in oncological conditions. VR-COG enhances learning and skill acquisition with better ecological efficiency than traditional cognitive remediation programs. VR approaches are well-received by oncology patients and show promise in reducing anxiety and depressive symptoms.

The trial aims to evaluate the effectiveness of highly specialized, nonpharmacological interventions on depressive symptoms and quality of life in oncology patients. Specifically, repetitive Transcranial Magnetic Stimulation (rTMS) and Virtual Reality-based Cognitive Remediation (VR-COG) will be analyzed, alongside standard Treatment as Usual (TAU), in comparison to TAU alone. This trial also aims at evaluate cognitive functioning, depression-related conditions and the cost-effectiveness of the interventions under study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of oncological disease in the last 5 years
* Diagnosis of Major Depressive Disorder, without psychotic symptoms, according to DSM-5 criteria
* 17-item Hamilton Rating Scale for Depression (HAM-D-17) (score ≥14)
* Age: 18 years or older
* Oncological disease in a non-advanced stage (Karnofsky Performance Status > 80)

Exclusion Criteria:

* Current or prior hospitalization in the next 6 months
* Planned surgery in the next 6 months
* Suicidal ideation
* Substance use
* History of significant head trauma, neurological disorders, intellectual deficits
* Recurrent seizures resulting from head trauma or conditions lowering seizure threshold
* Concurrent use of medications that increase the risk of epileptic seizures (e.g., antipsychotics, tricyclics, theophylline)
* Glaucoma, retinal detachment, or other serious vision impairments that may prevent the use of virtual reality technology
* Severe problems with autonomous ambulation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression rating scale (HAM-D 17) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  The Ham-D is the most widely used clinician-administered depression assessment scale.The original version contains 17 items pertaining to symptoms of depression experienced over the past week.
Dropout rates; Proportion of recruited participants among those considered eligible | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Feasibility will be assessed based on tolerability (dropout rates) and acceptability (proportion of recruited participants among those considered eligible).
Simulator Sickness Questionnaire (SSQ) | T0 (0 months - baseline); T1 (3 months - post intervention)
  Feasibility will be assessed based on side effects through Simulator Sickness Questionnaire (SSQ) self-report questionnaire that evaluates the frequency of unwanted effects due to virtual reality technologies, such as nausea, dizziness, headaches, eye strain, etc. 16 items.
TMSens_Q | T0 (0 months - baseline); T1 (3 months - post intervention)
  It was developed to report secondary effects following rTMS application. The use of the structured rTMS questionnaire will help to monitor the safety of rTMS.

SECONDARY OUTCOMES:
EuroQol (EQ)-5D | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is self-report questionnaire to assess quality of life and heath status according to five dimensions.
SF-12 | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a self-report questionnaire to assess quality of life considering two dimensions, about physical health and mental health.
Demoralization Scale (DS) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a 24-item self-administered questionnaire with four subscales: discouragement, loss of meaning/purpose, dysphoria, sense of failure.
Post-Traumatic Embitterment Disorder Self-Rating Scale | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a rating scale to assess embitterment reactions to negative life events
Brief Symptom Inventory (BSI) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Il is a questionnaire to evaluate symptoms of psychological distress
Insomnia Severity Index (ISI) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a tool to assess the severity of daytime and nighttime components of insomnia.
Biological Rhythms Interview for Assessment in Neuropsychiatry (BRIAN) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a scale consisting of 18 items to assess four areas of circadian rhythm difficulties: sleep, activity, social rhythms, and eating patterns.
Activities of Daily Living (ADL) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is an instrument to assess disability levels.
Psychosocial Adjustment to Illness (PAIS) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  I is a self-report instrument to assess seven dimensions about disability and quality of life.
Toronto Alexithymia Scale 20-item (TAS-20) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is a self-report questionnaire to assess alexithymia.
Screen for Cognitive Impairment in Psychiatry (SCIP) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  It is an instrument to assess cognitive deficit according to five subscales: immediate memory, working memory, phonemic verbal fluency, delayed memory, and psychomotor speed.
Trail Making Test | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Preliminary measures of effectiveness on executive function
Digit Span | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Preliminary measures of effectiveness on memory
Stroop Test | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Preliminary measures of effectiveness on executive function
Frontal Assessment Battery (FAB) | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Preliminary measures of effectiveness on executive function
Rey's Word Test | T0 (0 months - baseline); T1 (3 months - post intervention); T2 (3 months after T1); T3 (6 months after T1)
  Preliminary measures of effectiveness on memory
Matrix test | T0 (0 months-baseline), T1 (3 months - post intervention), T2 (3 months after T1), T3 (6 months after T1)
  Preliminary measure of effectiveness on selective attention.

OTHER OUTCOMES:
Cost-effectiveness | T0 (0 months - baseline); T3 (6 months after T1-post intervention)
  The cost effectiveness will be computed as the ratio of total costs divided by the mean improvements of quality of life across interventions (TAU, TAU+rTMS, TAU+VRCOG).
  Total costs will include the costs of the healthcare consultations (visits in the TAU condition), psychotropic drugs, equipment and staff.
  Total costs will be computed as the sum of these costs of each intervention, divided by the number of patients.
  Quality of life improvements will be computed as the difference between baseline (T0) vs endpoint (T3) quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Grassi, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (2):
- Italy (2):
  - Health Trust, Ferrara, Ferrara, FE
  - University Hospital of Cagliari, Cagliari